CLINICAL TRIAL: NCT06269926
Title: Cognitive Behavioral Therapy for Chronic Pain in Adults With Cerebral Palsy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Eric Chin, Assistant Professor of Neurology and Pediatrics, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00446666
Record Dates: First submitted 2024-02-13; First posted 2024-02-21 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-02

CONDITIONS: Cerebral Palsy; Pain, Chronic
Keywords: cerebral palsy; chronic pain; cognitive behavioral therapy; group therapy
MeSH Terms: conditions — Cerebral Palsy; Chronic Pain | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: The investigators will randomize 40 adults with cerebral palsy and pain-related impairment in daily activities into two study arms: Group 1 (CBT_now) will receive Cognitive Behavioral Therapy for Chronic Pain (CBT-CP; the primary intervention-a once weekly, 12-week group therapy course) shortly after enrollment. Group 2 (CBT_later) will receive CBT-CP after a three month delay. To maintain reasonable therapy cohort sizes (n=10 per cohort), each group (n=20 participants) will consist of two separate therapy cohorts (n=10 each). Participants will be evaluated at the beginning of the study, and then once every 3 months during the 12-month duration of the study.
Who Masked: Investigator
Masking Description: The team member responsible for efficacy analysis will be blinded to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT_later (Experimental): The CBT_later group will receive Cognitive Behavioral Therapy for Chronic Pain (CBT-CP; the primary intervention-a 12-week group therapy course) beginning approximately 3 months after enrollment.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Chronic Pain
- CBT_now (Experimental): The CBT_now group will receive Cognitive Behavioral Therapy for Chronic Pain (CBT-CP; the primary intervention-a 12-week group therapy course) beginning shortly after enrollment.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Chronic Pain

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Chronic Pain — CBT-CP consists of skill-based therapy sessions completed weekly for 12 weeks. Participants are oriented to CBT and set individualized goals (sessions #1-3) before focusing on cognitive and behavior skill building including physical activity, pacing, relaxation training, and cognitive restructuring (#4-10) then focusing on maintenance and discharge planning (#11-12). It will be completed in Maryland in an online real-time audio/video virtual group therapy format.

SUMMARY:
The purpose of this study is to understand if cognitive behavioral therapy can feasibly be provided to groups of adults with cerebral palsy and chronic pain via virtual group therapy sessions.

DETAILED DESCRIPTION:
Many adults with cerebral palsy have chronic pain that interferes with daily activities, but evidence regarding pain treatments for adults with cerebral palsy is limited. In other chronic pain patient populations, behavioral therapies such as cognitive behavioral therapy for chronic pain (CBT-CP) are a key component of evidence-based pain management. This study will assess challenges, implementation barriers, and preliminary efficacy of CBT-CP administered in a virtual group setting for adults with CP to design larger trials to definitively estimate treatment efficacy.

This study will invite 40 adult participants with CP and chronic pain that impacts their life to participate in a trial of CBT-CP. CBT-CP involves weekly group-therapy sessions for 12 weeks. Participants are oriented to CBT and set individualized goals (sessions #1-3) before focusing on cognitive and behavior skill building including physical activity, pacing, relaxation training, and cognitive restructuring (#4-10) then focusing on maintenance and discharge planning (#11-12). Participants will complete surveys every 3 months over a period of 12 months (a total of five surveys before and after CBT-CP). Participants will also continue to receive their usual medical care throughout.

All enrolled participants will receive the CBT intervention. Participants will be randomly assigned to receive CBT either upon enrollment (group 1; CBT_now) or after a three month delay (group 2; CBT_later).

This study will be conducted at the Kennedy Krieger Institute in Baltimore, Maryland, USA. Group CBT-CP will be conducted virtually via Zoom. 40 individuals with cerebral palsy who meet all inclusion/exclusion criteria will be recruited in two waves (one in early 2025 and one in early 2026). Participants must be at least 18 years old, able to make informed medical decision for themselves, and must endorse the ability and willingness to participate in all assessment and group sessions regardless of randomization outcome. Participants must also either live in Maryland, or be able to travel to Maryland on a weekly basis for the group therapy sessions.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. Has a diagnosis of cerebral palsy
3. Able to send and receive information effectively with familiar communication partners
4. Able, during the consent process, to answer questions about the study to indicate that they understand and consent to participation
5. Has pain that at least moderately interferes with some aspect(s) of their daily activities
6. Able and willing to participate in all assessment and group sessions regardless of randomization outcome
7. Appears on a screening assessment to have enough cognitive ability to recognize their thoughts, feelings, and behaviors to be able to benefit from CBT-CP

Exclusion Criteria: (if met then participant will not eligible to participate)

1. Previously received Cognitive Behavioral Therapy (CBT) for chronic pain
2. Endorses that most of their pain is attributable to a recent event (e.g. trauma, surgery that occurred in the past 3 months)
3. Unable to attend weekly CBT-CP sessions from a location in the state of Maryland

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2025-02-27 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Data collection achieved (feasibility assessment) | Five assessments (at enrollment and at 3, 6, 9, and 12 months post-enrollment)
  We will examine the rate of survey completion for each survey (0 = survey incomplete, 1 = survey complete). Higher scores indicate a better outcome (greater feasibility of recruiting adults with CP and chronic pain and retaining their engagement to complete this clinical trial over a period of 12 months).

SECONDARY OUTCOMES:
Therapy attendance | Weekly x 12 weeks during therapy administration
  Therapists will track frequency of group therapy attendance (present/absent) for each participant throughout the 12 week intervention. We will assess the rate of treatment adherence by looking at the number of sessions attended by each participant over the course of the intervention, as well as at a cohort level
Patient Global Impressions of Change | Four assessments (at 3, 6, 9, and 12 months post-enrollment)
  These questions ask about how participants feel now, compared to before the intervention. Responses are recorded on a 7-point scale ranging 1 being "very much worse" to 7 being "very much improved"; higher scores represent better outcomes.
Change in Pain Catastrophizing Scale score | Will be assessed at baseline (prior to randomization) as well as every 3 months throughout the 12 month study timeframe for each cohort
  The Pain Catastrophizing Scale assesses specific patterns of pain-related thoughts. Responses are recorded on a 5-point scale, with 1 being "Not at all" and 5 being "All the time". Higher scores represent worse outcomes.
Change in Pain Self-Efficacy-4 Score | Will be assessed at baseline (prior to randomization) as well as every 3 months throughout the 12 month study timeframe for each cohort
  This 4-item questionnaire assesses an individual's confidence in their ability to complete various activities despite the presence of pain. Responses are recorded on a 7-point scale, with 1 being "Not at all confident" and 7 being "Completely confident". Higher scores represent better outcomes.
Changes in Brief Pain Inventory Pain Interference Subtest scores | Will be assessed at baseline (prior to randomization) as well as every 3 months throughout the 12 month study timeframe for each cohort
  This survey asks how much pain is interfering with various activities. Responses are recorded on a 10-point scale, with 1 being "Does not interfere" and 7 being "Completely interferes". Higher scores represent worse outcomes. We will examine 1) improvement in the activity that saw the greatest pain-related impairment at baseline and 2) average improvement across all activities listed.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Intensity 3a T-score | Will be assessed at baseline (prior to randomization) as well as every 3 months throughout the 12 month study timeframe for each cohort
  These questions ask about pain levels over the previous 7 days. Responses are recorded on a 5-point scale, with 1 being "had no pain" and 5 being "very severe"; higher scores represent worse outcomes.
Changes in Patient Health Questionnaire-4 (PHQ-4) | Will be assessed at baseline (prior to randomization) as well as every 3 months throughout the 12 month study timeframe for each cohort
  This 4-item questionnaire asks about symptoms of anxiety and depression in the last 14 days. Responses are recorded 4-point scale, with 0 being "not at all" and 4 being "nearly every day"; higher scores represent worse outcomes. We will examine changes in anxiety symptom scores and in depression symptom scores.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Chin, M.D, Principal Investigator — Kennedy Krieger Institute, Johns Hopkins University
Locations (1):
- Kennedy Krieger Institute, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No